CLINICAL TRIAL: NCT02371382
Title: Multicentre Prospective Study to Evaluate Long-term Clinical Outcomes of the Sirius Cemented Femoral Stem
Acronym: Sirius
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.H41
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Arthroplasty, Replacement, Hip
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Arthroplasty hip — Hip replacement

SUMMARY:
The purpose of this multicentre, prospective study is:

* Document the Clinical and Radiographic performance of the stem at 3 months, 1 year, 3 years, 5 years, 7 and 10 years.
* Report Safety and Survivorship up to 10 years F/up.

DETAILED DESCRIPTION:
This study intends to evaluate the safety and performance of the Sirus cemented hip stem in terms of function improvement postoperatively, stability and fixation of femoral stem and survivorship.

ELIGIBILITY:
Inclusion Criteria:

Selection of subjects for this evaluation should be in accordance with the indications of Sirus stem:

1. Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
2. Rheumatoid arthritis
3. Correction of functional deformity
4. Treatment of non-union, femoral neck fracture and trochanteric fractures of the proximal femur with head involvement, unmanageable using other techniques.
5. Revision procedures where other treatments or devices have failed. The Sirius Femoral Hip Stem is intended for cemented use only and may be used in partial and total hip arthroplasties

Exclusion Criteria:

* Absolute contraindications include:

infection, sepsis, osteomyelitis

Additional contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* Osteoporosis,
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy or neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: minimum age: 18 maximum age: gender: both
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-03; Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 1 year
  Change in Harris Hip Score from Baseline to 1 Year post-surgery, Harris Hip Score, 0-100 points. The higher the positive difference between baseline and follow up the better the result

SECONDARY OUTCOMES:
Oxford Hip score | 10 years
  Oxford Hip Score at 1,3,5, 7 and 10 year postop, Oxford Hip score 0-48 points, The higher the positive difference the better the result.

CONTACTS AND LOCATIONS:
Overall Officials: Alun John, Principal Investigator — University Hospital of Wales; Per Kjærsgaard-Andersen, MD, Principal Investigator — Lillebaelt Hospital Vejle, Denmark
Locations (2):
- Sygehus Vejle, Vejle, Denmark
- University Hospital of Wales, Llandough Hospital, Penarth, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No